CLINICAL TRIAL: NCT00592540
Title: Unrelated Donor Bone Marrow Transplantation for Definitive Treatment of Patients With Phosphoglycerate Kinase (PGK) Deficiency
Brief Title: Unrelated Donor BMT for Treatment of Patients With PGK Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060486
Record Dates: First submitted 2007-12-26; First posted 2008-01-14 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Phosphoglycerate Kinase (PGK) Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unrelated Donor BMT (Experimental)
  Interventions: Procedure: Unrelated Donor BMT

INTERVENTIONS:
Procedure: Unrelated Donor BMT — Unrelated donor bone marrow transplantation has not been performed with these patients in the past

SUMMARY:
Phosphoglycerate kinase (PGK) deficiency is a rare x-linked disorder characterized by hemolytic anemia, seizures, muscle fatigue, and progressive neurological dysfunction. The disease is caused by the deficiency of PGK, an enzyme required for ATP formation through the glycolytic pathway. PGK is an enzyme that is ubiquitous to all cells of the human body, but red blood cells, muscles, and nerve cells are most severely affected by the absence of PGK due to their reliance upon the glycolytic pathway. Mutations of the PGK gene are highly variable and result in diverse phenotypes, ranging from mild hemolytic anemia only to severe mental retardation and early death in childhood. The more severe phenotypes show progressive neurologic deterioration between infancy and adolescence.

This is a 2 patient study aimed at studying the role of stem cell transplant in PGK deficiency. Because the disease is so rare, the study will be limited to the 2 sibling patients followed by our group, though it would be open to other participants who would meet inclusion/exclusion criteria if such presented to us. The objective of this study is to evaluate the feasibility and efficacy of stem cell transplants to treat patients with PGK deficiency, Amiens subtype.

DETAILED DESCRIPTION:
Phosphoglycerate kinase (PGK) deficiency is a rare x-linked disorder characterized by hemolytic anemia, seizures, muscle fatigue, and progressive neurological dysfunction. The disease is caused by the deficiency of PGK, an enzyme required for ATP formation through the glycolytic pathway. PGK is an enzyme that is ubiquitous to all cells of the human body, but red blood cells, muscles, and nerve cells are most severely affected by the absence of PGK due to their reliance upon the glycolytic pathway. Mutations of the PGK gene are highly variable and result in diverse phenotypes, ranging from mild hemolytic anemia only1 to severe mental retardation and early death in childhood.2-5 The more severe phenotypes show progressive neurologic deterioration between infancy and adolescence.2,3,5 PGK-Amiens refers to a particular mutation that is an A to T transversion, which predicts an amino acid change of aspartate (Asp: GAT) to valine (Val: GTT) at the 164th position from the NH2-terminal methionine residue. This D164V mutation has been identified previously as PGK-Amiens or PGK-New York in a French and in a Chinese family respectively.3,6 This particular mutation results in the most severe phenotype. All 6 of the boys described in the literature with this mutation have had progressive neurologic decline, seizures, episodes of hemiplegia, aphasia, emotional lability, and severe hemolytic crises. Two of the boys died in childhood, 2 are institutionalized with no ability to communicate or provide self-care, and 2 are moderately mentally retarded with seizures and hemolytic anemia. The two brothers cared for at this institution have the Amiens variant of PGK deficiency.

Allogeneic bone marrow transplantation (BMT) became feasible in the 1960s after elucidation of the Human Leukocyte Antigen (HLA) complex. Since then, the therapy has evolved into an effective therapy for many hematologic disorders(7). Otherwise incurable malignancies are frequently cured by this approach, with the likelihood of cure ranging from 10% to 85%, depending on the disease and disease-status. The treatment strategy incorporates very large doses of chemotherapy and often radiation to eliminate malignant cells and to immunosuppress the recipient enough to allow engraftment of donor cells. Donor cells give rise to hematopoiesis within two to three weeks, rescuing the patient from the effects of high dose therapy. In the ideal circumstance, immune recovery and recipient-specific tolerance occurs over the following 6-18 months, and the patient is cured of his or her underlying hematologic disorder, off of immunosuppression, with a functionally intact donor-derived immune system. However, complications of the process are common and include potentially permanent or fatal organ damage from the effects of high dose chemotherapy, infection, hemorrhage, and, in particular, graft-versus-host-disease. A realistic estimate of transplant-related mortality, including deaths due to acute and chronic graft-versus-host diseases, in the standard HLA-matched sibling setting is as high as 25%. The risk of treatment related mortality thus limits the success of the approach even in younger patients and certainly precludes its use in older patients. Thus, particularly for older patients, new strategies in transplantation are needed.

Stem cells for allogeneic transplant are traditionally obtained from one of three sources: bone marrow (1), peripheral blood stem cells mobilized by provision of the growth factor GCSF (2), or umbilical cord blood (3). Each source has specific advantages and disadvantages. The desired source of stem cells for allogeneic transplant is a matched sibling donor. However, if that is not feasible, a matched unrelated donor can be sought through the National Marrow Donor Program (NMDP). The National Marrow Donor Program (NMDP) in Minneapolis, Minnesota, was established in 1986 to facilitate the search for, and procurement of, HLA-matched marrow from volunteer, unrelated marrow donors for patients with life-threatening diseases curable by SCT (7). The NMDP network consists of 99 donor centers, 108 collection centers, 150 transplant centers and a Coordinating Center in Minneapolis. As of June 29, 2003, the NMDP had a registry of 5,032,382 volunteer marrow donors and 28,574 cord blood units stored, and had facilitated 13,213 unrelated marrow transplants (marrow, PBSC and cord blood) worldwide. Over 600,000 donors in the NMDP Registry are contributed by European registries, which are affiliated with the NMDP. In addition, approximately 1 million donors are available by searching NMDP International Cooperative Registries in Europe, South America, and Asia. On average, searching patients have a 75% chance of finding a match within the NMDP, with a median time from search to transplant of less than 6 months. Vanderbilt University Medical Center is a NMDP approved aphaeresis center, collection center and transplant center and adheres to the policies and procedures of the NMDP as outlined in The 18th Edition of the NMDP Standards (effective since September 13th, 2002, implemented February 10th, 2003).

Stem cell transplantation (SCT) has been performed in children with various metabolic diseases, including mucopolysaccharide disorders (MPS), leukodystrophies, and glycoprotein metabolic disorders.8 The prototypical metabolic disorder for SCT is Hurler syndrome, or MPS IH. Hurler syndrome results from the lack of a lysosomal enzyme needed to degrade glycosaminoglycans, which then build up and cause progressive intellectual decline, hepatosplenomegaly, cardiac valvular disease, airway abnormalities, and skeletal abnormalities. SCT performed early in the disease process leads to enzyme replacement and stops progression of disease.9 SCT has helped other MPS disorders including severe Maroteaux-Lamy syndrome and Sly syndrome, but unfortunately, and for reasons not well understood, SCT has not helped in several other MPS disorders, such as Hunter, Sanfilippo, and Morquio syndromes.8 X-linked adrenoleukodystrophy is a disease that affects boys with variable degrees of severity. When boys show early MRI changes and undergo SCT, outcome is very good, with preservation of neurological and neurocognitive function.10,11 Other leukodystrophies that respond to early SCT include Krabbe disease and metachromatic leukodystrophy.8,12 Glycoprotein metabolic disorders are exceedingly rare and thus there is limited experience with SCT in patients with these disorders. There have been successful outcomes in preservation of cognitive function in α-mannosidosis,13 fucosidosis,14 Batten disease,15 and Gaucher disease Type I.16 SCT has not been able to salvage children with Fabry disease, Tay Sachs disease, Pompe disease, and Sandhoff disease.8 Again, it is poorly understood why SCT is able to stop neurologic decline in some metabolic disorders and not others.

Definitive therapy for PGK deficiency necessarily involves production of the PGK enzyme. The hemolytic anemia that is part of this disease could be cured by allogeneic stem cell transplant, as replacing the hematopoietic system would ensure production of the enzyme in the red blood cells. However, the neurologic complications of the disease would require that the enzyme can find its way into the neurons themselves. Because of the rarity of PGK deficiency, there has been as yet no controlled study to define the most efficacious approach. In fact, there is no mention of any therapy in the literature. There is currently no enzyme replacement therapy and no major research effort underway to do so. To our knowledge, stem cell transplant in this disease has not been performed except for in one 7 month old child with PGK-Amiens in Australia, who is currently being prepared for SCT. The stem cell source will be determined by the donor availability. The donor registry allows the donor the option of donating either peripheral blood or bone marrow.

(Please note all reference numbers refer to the Reference list of the study protocol, pages 9 and 10.)

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender and between 3 and 12 years of age.
* Patients diagnosed with PGK deficiency.

Exclusion Criteria:

* Patients must have organ function (heart, lung, kidney, liver) that is sufficient for bone marrow transplant, determined by the standard of care for allogeneic bone marrow transplant.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2006-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and efficacy of stem cell transplants to treat two patients with PGK deficiency, Amiens subtype. | 5+ years

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M. Rhodes, MD, Principal Investigator — Vanderbilt Children's Hospital
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Background] Lake BD, Steward CG, Oakhill A, Wilson J, Perham TG. Bone marrow transplantation in late infantile Batten disease and juvenile Batten disease. Neuropediatrics. 1997 Feb;28(1):80-1. doi: 10.1055/s-2007-973677. PMID 9151332
- [Background] Miano M, Lanino E, Gatti R, Morreale G, Fondelli P, Celle ME, Stroppiano M, Crescenzi F, Dini G. Four year follow-up of a case of fucosidosis treated with unrelated donor bone marrow transplantation. Bone Marrow Transplant. 2001 Apr;27(7):747-51. doi: 10.1038/sj.bmt.1702994. PMID 11360116
- [Background] Shapiro E, Krivit W, Lockman L, Jambaque I, Peters C, Cowan M, Harris R, Blanche S, Bordigoni P, Loes D, Ziegler R, Crittenden M, Ris D, Berg B, Cox C, Moser H, Fischer A, Aubourg P. Long-term effect of bone-marrow transplantation for childhood-onset cerebral X-linked adrenoleukodystrophy. Lancet. 2000 Aug 26;356(9231):713-8. doi: 10.1016/S0140-6736(00)02629-5. PMID 11085690
- [Background] Peters C, Shapiro EG, Anderson J, Henslee-Downey PJ, Klemperer MR, Cowan MJ, Saunders EF, deAlarcon PA, Twist C, Nachman JB, Hale GA, Harris RE, Rozans MK, Kurtzberg J, Grayson GH, Williams TE, Lenarsky C, Wagner JE, Krivit W. Hurler syndrome: II. Outcome of HLA-genotypically identical sibling and HLA-haploidentical related donor bone marrow transplantation in fifty-four children. The Storage Disease Collaborative Study Group. Blood. 1998 Apr 1;91(7):2601-8. PMID 9516162
- [Background] Peters C, Steward CG; National Marrow Donor Program; International Bone Marrow Transplant Registry; Working Party on Inborn Errors, European Bone Marrow Transplant Group. Hematopoietic cell transplantation for inherited metabolic diseases: an overview of outcomes and practice guidelines. Bone Marrow Transplant. 2003 Feb;31(4):229-39. doi: 10.1038/sj.bmt.1703839. PMID 12621457
- [Background] Cosentino M, Bombelli R, Ferrari M, Marino F, Rasini E, Maestroni GJ, Conti A, Boveri M, Lecchini S, Frigo G. HPLC-ED measurement of endogenous catecholamines in human immune cells and hematopoietic cell lines. Life Sci. 2000 Dec 8;68(3):283-95. doi: 10.1016/s0024-3205(00)00937-1. PMID 11191644
- [Background] Cohen-Solal M, Valentin C, Plassa F, Guillemin G, Danze F, Jaisson F, Rosa R. Identification of new mutations in two phosphoglycerate kinase (PGK) variants expressing different clinical syndromes: PGK Creteil and PGK Amiens. Blood. 1994 Aug 1;84(3):898-903. PMID 8043870
- [Background] Noel N, Flanagan JM, Ramirez Bajo MJ, Kalko SG, Manu Mdel M, Garcia Fuster JL, Perez de la Ossa P, Carreras J, Beutler E, Vives Corrons JL. Two new phosphoglycerate kinase mutations associated with chronic haemolytic anaemia and neurological dysfunction in two patients from Spain. Br J Haematol. 2006 Feb;132(4):523-9. doi: 10.1111/j.1365-2141.2005.05882.x. PMID 16412025
- [Background] Valentine WN, Hsieh HS, Paglia DE, Anderson HM, Baughan MA, Jaffe ER, Garson OM. Hereditary hemolytic anemia: association with phosphoglycerate kinase deficiency in erythrocytes and leukocytes. Trans Assoc Am Physicians. 1968;81:49-65. No abstract available. PMID 5721411